CLINICAL TRIAL: NCT00110539
Title: Internet-Based Curriculum About Herbs and Dietary Supplements
Brief Title: Effectiveness of an Internet-Based Curriculum in Increasing Health Care Providers' Knowledge of Herbs and Dietary Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Library of Medicine (NLM) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: R01LM007709 (NIH)
Record Dates: First submitted 2005-05-10; First posted 2005-05-11 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2006-08

CONDITIONS: Healthy
Keywords: Medicine, Herbal; Dietary Supplements; Complementary and Alternative Medicine; Physicians

INTERVENTIONS:
Behavioral: Complementary and alternative medicine education

SUMMARY:
The purpose of this study is to determine the effectiveness of four different strategies designed to improve clinicians' knowledge about herbs and dietary supplements. This study will also increase their confidence in their ability to answer patient questions about these topics.

Study hypotheses: 1) Delivery of modules over 10 weeks will lead to better educational outcomes than delivery of modules at one time. 2) The method of module delivery that directly lists the modules in an email will be associated with greater improvements in knowledge, confidence, and communication skills and greater satisfaction with the overall curriculum than methods that involve the delivery of only links to the modules in an email. 3) Active participation in a moderated mailing list will enhance outcomes and satisfaction with the curriculum more than non-participation or passive participation (reading the messages of others). 4) More positive attitudes toward the use of and greater use of computer and Internet technologies at baseline will be associated with more active participation in the mailing list; greater use of the modules delivered through links; greater improvements in knowledge, confidence, and communication; and more positive attitudes about the curriculum following participation in the study.

DETAILED DESCRIPTION:
As herbal medicine use becomes more popular, health care providers may find that patients are asking questions about the risks and benefits of complementary and alternative medicine (CAM) more frequently. It is important that providers have some knowledge about these therapies and are familiar with resources to which they can refer patients. This study will compare the effectiveness of four strategies used to deliver educational modules that can increase health care providers' knowledge about herbal medicine and dietary supplements.

This study will last about 10 weeks and will enroll a variety of health care providers, including physicians, physician assistants, pharmacists, dietitians, and nurses. At study entry, participants will be stratified by provider type. Participants will then be randomly assigned to 1 of 4 educational delivery strategies: delivery of educational modules all at one time directly through email, delivery of modules over 10 weeks directly through email, delivery of modules through an email message with a link to an Internet site containing all modules, or delivery of multiple emails over 10 weeks with links to an Internet site containing all modules.

Each module will begin with a brief clinical scenario followed by questions to assess knowledge, confidence about where to locate information, and the level of communication that providers have engaged in with their patients. Participants will complete questionnaires at study entry and at Week 10. The questionnaires will assess the use of and attitudes toward Internet technology, motivation for participating in the course, and knowledge, attitudes, and communication practices related to the clinical use of herbs and dietary supplements. Participants will have the opportunity to participate in a moderated mailing list where they can discuss CAM-related topics with other providers and read the discussions of others. In addition, after completing the curriculum, participants will complete questionnaires about their use of and attitudes toward the intervention they received in the study.

ELIGIBILITY:
Inclusion Criteria:

* Live and work in the United States
* Licensed to provide health care in the United States
* Have regular access to the Internet and an e-mail address that can be checked at least twice weekly for at least 4 months
* Willing to complete all study assessments

Exclusion Criteria:

* Previous enrollment in this curriculum

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 2004-02; Study Completion 2004-12

PRIMARY OUTCOMES:
Changes in participant knowledge, confidence, and communication practices regarding herbs and dietary supplements

SECONDARY OUTCOMES:
Impact of comfort with using technology on the primary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Kathi Kemper, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Northwest Area Health Education Center, Winston-Salem, North Carolina, United States